CLINICAL TRIAL: NCT06554262
Title: Optimal Visceral Fat Area Cutoffs for Screening Cardiometabolic Risk: a Large-scale Population-based Cohort Study
Brief Title: Visceral Fat and Cardiometabolic Risk
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Xia Wang, Principal Investigator, Capital Medical University
Other Study IDs: 2012062
Record Dates: First submitted 2024-08-10; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Cardiometabolic Risk; Visceral Fat; Cohort Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiometabolic risk group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was involved in this study

SUMMARY:
The present study showed that the 75th percentile of visceral fat area in boys and girls is the optimal cutoff for screening cardiometabolic risk and its clustering, but the 80th percentile is the optimal cutoff for hyperglycemia screening in girls. The investigators proposed simplified cutoffs of 37.19 cm2 and 31.09 cm2 aged 6 to 8 years, 56.76 cm2 and 39.51 cm2 aged 9 to 11 years, 57.03 cm2 and 38.33 cm2 aged 12 to 15 years, and 58.32 cm2 and 53.91 cm2 aged 16 to 18 years for boys and girls, respectively. Both the optimal and simplified methods were verified in a 2-year longitudinal cohort. An improved understanding of the importance of visceral fat to cardiometabolic risk and its clustering in children may yield insight into the risks associated with child obesity and the initial phases of cardiovascular disease development, especially in normal-weight boys.

ELIGIBILITY:
Inclusion Criteria:

Healthy children and adolescents aged 6-18 years

Exclusion Criteria:

Heart disease Kidney disease Thyroid disease Individuals who take hormone medication Missing data for anthropometry

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: A total of 8133 participants (mean age =11.8 years, SD =3.3 years) from the China Child and Adolescent Cardiovascular Health completed the visceral fat area assessment by dual-energy X-ray absorptiometry, and 10805 participants from the school-based cardiovascular and bone health program (mean age =11.0 years, SD =3.3 years).
Sampling Method: Non-Probability Sample
Enrollment: 18938 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Visceral fat area cutoffs and cardiometabolic risk | 2 years
  Based on dual-energy X-ray measurements of visceral fat area, age- and sex-specific visceral fat area cutoffs for screening cardiometabolic risk was developed and validated.